CLINICAL TRIAL: NCT05915065
Title: Intuitively Controlled Virtual Reality to Treat Phantom Limb Pain
Brief Title: VR to Evaluate Phantom Limb Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Coapt, LLC (Industry)
Responsible Party: Principal Investigator, Levi Hargrove, Scientific Chair, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00213205
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Phantom Limb Pain; Phantom Pain; Phantom Sensation; Phantom Limb Syndrome With Pain; Phantom Pain Following Amputation of Lower Limb; Phantom Pain Following Amputation of Upper Limb; Amputation; Upper Limb Amputation at the Hand; Upper Limb Amputation at the Wrist; Upper Limb Amputation Below Elbow (Injury); Upper Limb Amputation Above Elbow (Injury); Lower Limb Amputation Knee; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Below Knee (Injury); Lower Limb Amputation at Ankle (Injury)
Keywords: Virtual Reality; Limb Loss; Amputation; Phantom Pain
MeSH Terms: conditions — Phantom Limb; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This study will enroll one, non-random group of amputees to participate in 2-4 in person or virtual research visits, participate in a home trial and complete questionnaires pre home trial, at various points during the home trial and upon conclusion of the home trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phantom Limb Pain Management System during at-home use. (Other): Participants attend either in person at Shirley Ryan AbilityLab or virtually via Zoom
  * Educational documents provided on pain and phantom limb pain.
  * Participants are measured for an electrode cuff either in person or virtually
  * Complete several questionnaires.
  * Provided training on the Phantom Limb Pain Program with use of the electrode cuff and muscular contractions of their limb
  * Participate in a 8 week home trial (1.5 hours per week of use, 20-40 minutes, 4-5x each week)
  * Once home trial is complete - participants will be asked to participate in a phone or Zoom call at weeks 16,24 and 32 to repeat questionnaires.
  Interventions: Device: Coapt Phantom Limb Pain Management System

INTERVENTIONS:
Device: Coapt Phantom Limb Pain Management System — The PLP-MS consists of (1) an expandable arm/leg cuff with electrode sensors to collect EMG signals from residual limb muscles, (2) an integrated hardware module (the Coapt Complete Control Gen2.5 system) that translates users' EMG signals into game commands, (3) game software for mobile applications, and (4) a secure, HIPAA-compliant cloud-based data storage system for storing and retrieving user data remotely.

SUMMARY:
The objective of this study is to develop a virtual rehabilitation system that can be used to effectively treat Phantom Limb Pain (PLP) within the research setting and for at-home use by individuals with upper and lower extremity amputation.

We hypothesize that the system will improve PLP for individuals with upper or lower extremity amputation, as measured through with various outcome measures and questionnaires.

DETAILED DESCRIPTION:
The objective of this study is to develop a virtual rehabilitation system that can be used to effectively treat Phantom Limb Pain (PLP) within the research setting and for at-home use by individuals with upper and lower extremity limb absence.

Phase 1: Complete in-lab or virtual iterative usability and functionality testing of hardware and software components of The Coapt Phantom Limb Pain Management System to ensure readiness for at-home use - COMPLETED

Phase 2: A clinical trial of The Coapt Phantom Limb Pain Management System during at-home use. We hypothesize that the system will improve PLP for individuals with upper or lower extremity absence, as measured through various questionnaires.

VR systems have been proposed as alternative technologies to treat PLP since they are relatively inexpensive and more readily available. Virtual reality environments allow for real-time control practice utilizing different tasks and games, and have been widely accepted as clinically viable options for administering therapy.

Effective PLP treatment methods are needed for individuals with limb absence that can be utilized on an as-needed basis in the home. VR therapy could potentially be an effective treatment for individuals with chronic upper or lower limb PLP.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years old
* Amputation of the upper or lower limb, including amputation of multiple limbs
* English Speaking
* Chronic phantom limb pain (at least 6-months duration)
* Average phantom limb pain intensity of 4 or greater on a 0-10 numerical rating scale
* Average frequency of phantom limb pain episode of at least twice per month.
* Residual limb pain of less than 5 on the Numerical Pain Rating Scale
* Pain medication use stable for > 1 month

Exclusion Criteria

* Unable to tolerate use of liner or cuff on their residual limb
* Skin irritation/wounds on residual limb that would prevent use of the electrode cuff
* Significant cognitive deficits or visual impairment that would preclude them from giving informed consent or following instructions during the experiments, or the ability to obtain relevant user feedback.
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Short-form McGill Pain Questionnaire | Baseline score and at the post-treatment assessment at the end of the 8-week intervention
  The primary outcome measure in this study is change in the pain rating index (PRI) between the baseline score and at the post-treatment assessment at the end of the 8-week intervention. The PRI is computed as the sum of the scores for all descriptors of the Short Form of the McGill Pain Questionnaire (SF-MPQ).

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline score and at the post-treatment assessment at the end of the 8-week intervention
  The pain VAS is a unidimensional measure of pain intensity, used to record a persons pain progression, or compare pain severity between paints with similar conditions.
Numerical Pain Rating Scale (NPRS) | Baseline score and at the post-treatment assessment at the end of the 8-week intervention
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Patient-Reported Outcomes Measurement Information Systems (PROMIS) | Baseline score and at the post-treatment assessment at the end of the 8-week intervention
  ROMIS® (Patient-Reported Outcomes Measurement Information System®) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults. PROMIS measures can be used with the general population and with individuals living with chronic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States